CLINICAL TRIAL: NCT03025035
Title: Open Label, Phase II Pilot Study of Immune Checkpoint Inhibition With Pembrolizumab in Combination With PARP Inhibition With Olaparib in Advanced BRCA-mutated or HDR-defect Breast Cancers
Brief Title: Pembrolizumab in Combination With Olaparib in Advanced BRCA-mutated or HDR-defect Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuan Yuan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Yuan Yuan, Director, Breast Oncology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015-18-Mita-MK3475
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Results first posted 2025-05-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: BRCA-mutation; Immune checkpoint inhibition; Immunotherapy; Advanced BRCA-mutated breast cancer; HDR-defect; PARP inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Olaparib (Experimental): This is an open-label, single-arm pilot study of pembrolizumab (study drug) in combination with Olaparib in 20 subjects with advanced BRCA mutation or HDR-defect associated breast cancer having progressed through at least a standard first line therapy.
  Interventions: Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab IV solution administered on Day 1 of each 3-week cycle
  Other Names: Keytruda; MK-3475
Drug: Olaparib — Olaparib administered orally twice a day
  Other Names: Lynparza

SUMMARY:
This trial will evaluate the use of immunotherapy and PARP inhibition in a population with incurable advanced breast cancer associated with a germline BRCA mutation or HDR-defect. The main objective is to examine overall response rate of pembrolizumab (immunotherapy) in combination with Olaparib (PARP inhibitor) in advanced BRCA-mutated or Homology-directed repair (HDR)-defect breast cancer.

DETAILED DESCRIPTION:
There are two BRCA genes, BRCA1 and BRCA2, and they play a role in protecting cells from cancer. HDR-defect is another type of gene mutation that can contribute to development and progression of cancer. If one of these genes is mutated, cells may rapidly change and divide, which can lead to cancer. Pembrolizumab is a drug that works with the immune system to target the tumor (immunotherapy). The investigators want to know if combining pembrolizumab and Olaparib therapy will be able to reduce the size and amount of cancer cells with fewer side effects than standard treatment by targeting the tumor. This research study is designed to test the investigational use of pembrolizumab and Olaparib in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Be ≥18 years of age on day of signing informed consent
* Advanced BRCA-mutated and/or HDR-defect breast cancer progressing on or after prior therapy for metastatic disease or locally advanced disease; Prior therapy is defined as follows: for triple negative breast cancer - progressing after at least 1 line of any prior chemotherapy; for HER2 positive disease must have progressed after at least two HER2 directed therapies in the metastatic setting including ado-trastuzumab emtansine (T-DM1); for hormone receptor positive disease (ER, PR, or both) must have progressed after a CDK4/CDK6 inhibitor plus hormonal therapy. Patients with progression within 12 months from previous neoadjuvant or adjuvant treatment could be enrolled in the study as 1st line therapy in metastatic setting.
* Measurable disease by RECIST 1.1, with at least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements. Patients with non-measurable bone metastases in addition to measurable disease are eligible; however patients with non-measurable bone disease as the only site(s) of disease are not eligible.
* ECOG 0 or 1
* Documented BRCA deleterious germline or somatic mutation and/or HDR-defect.
* FFPE tumor tissue available for analysis
* Adequate organ function
* Female subjects: Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

  1. Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
  2. radiation-induced oophorectomy with last menses >1 year ago
  3. chemotherapy-induced menopause with >1 year interval since last menses
  4. surgical sterilization (bilateral oophorectomy or hysterectomy)
* Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination. This should be started from the signing of the informed consent and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse.
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential
* Patients must have a life expectancy ≥ 16 weeks

Exclusion Criteria:

* Is currently participating or has participated in a study of investigational agent or using an investigational device with 30 days of the first dose of pembrolizumab.

  1. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1.
  2. Subjects must have recovered (i.e., ≤ Grade 1 or at baseline) from any adverse events due to a previously administered agent. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  3. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Is receiving systemic steroid therapy within three days prior to the first dose of pembrolizumab or receiving any other form of immunosuppressive medication
* Is expected to require any other form of systemic or localized antineoplastic therapy while on trial.

  1. Subjects with ER+/PR+ disease may be given endocrine therapy.
  2. Subjects with HER2+ disease will be required to discontinue trastuzumab (Herceptin).
* Has participated in another MK03475 trial.

  a. Note: Patients with or without prior PARP-inhibitor exposure may be included.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Has known hypersensitivity to pembrolizumab or any of its excipients
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known history of prior malignancy except if the patient has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by MRI for at least four weeks prior to the first dose of pembrolizumab and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are using no steroids for at least three days prior to study medication.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has active tuberculosis
* Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of pembrolizumab. Administration of killed vaccines is allowed.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Subjects with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Subjects that require inhaled steroid or local steroid injections will not be excluded from the study. Subjects with hypothyroidism not from autoimmune disease and stable on hormone replacement will not be excluded from the study. Note: Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has had an allogenic tissue / solid organ transplant.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit (Visit 1) through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2025-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Olaparib: This is an open-label, single-arm pilot study of pembrolizumab (study drug) in combination with Olaparib in 20 subjects with advanced BRCA mutation and/or HDR-defect associated breast cancer having progressed through at least a standard first line therapy.
  Pembrolizumab: Pembrolizumab IV solution administered on Day 1 of each 3-week cycle
  Olaparib: Olaparib administered orally twice a day
Period: Overall Study
Arm/Group | Pembrolizumab + Olaparib
Started | 14
Completed | 11
Not Completed | 3
Not completed — Death | 2
Not completed — Disease progression and was taken off study. Only received pembrolizumab & is not evaluable. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Olaparib
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.45455 (13.09476)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per RECIST1.1
Description: Defined as complete or partial response or stable disease per RECIST 1.1 criteria with assessment every 9 weeks during the first year and while on the study drug, and every 12 weeks thereafter. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), a tumor that is neither shrinking sufficiently to be considered a partial response (PR) (at least 30% decrease in tumor burden), nor growing significantly enough to be considered progressive disease (PD) (more than 20% increase in tumor burden); Overall Response (OR) = CR + PR + SD
Time Frame: Up to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Olaparib
Number analyzed (Participants) | 11
Participants | 7

2. Secondary Outcome: Progression Free Survival (PFS), Per RECIST 1.1
Description: As measured by RECIST 1.1, in patients progressing after 1st line therapy
Time Frame: Up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival (OS)
Description: Calculated in months from the start of treatment to the date of death from any cause
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Benefit Rate (CBR = CR+PR+SD) Per RECIST 1.1
Description: As measured by RECIST 1.1, in patients progressing after 1st line therapy
Time Frame: Up to 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Duration of Response (DOR) for Complete Response (CR) and Partial Response (PR) Per RECIST 1.1
Description: As measured by RECIST 1.1, in patients progressing after 1st line therapy
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are collected for up to two years of total study participation.
Arm/Group | Pembrolizumab + Olaparib
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Olaparib (N=11)
Anemia Hemoglobin (Blood and lymphatic system disorders) | 6 (14)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 1 (1)
Concentration Impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Edema Limbs (General disorders) | 2 (2)
Eye disorders - Other (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eyelid Function Disorder (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 4 (4)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastroesophagael Reflux (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Non-Cardiac Chest Pain (General disorders) | 1 (2)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Other- Pain at Biopsy Site (General disorders) | 1 (1)
Other- Tinnitus (Ear and labyrinth disorders) | 1 (1)
Other- Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Cardiac disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
White blood cell decreased (Injury, poisoning and procedural complications) | 1 (1)
Other- Injection Site Pain (Intermittent) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT03025035/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03025035/ICF_001.pdf